CLINICAL TRIAL: NCT07112833
Title: A Phase II Clinical Study of Induction Adebrelimab Combined With Chemotherapy Followed by Concurrent Chemoradiotherapy for Locally Advanced Unresectable Esophageal Squamous Cell Carcinoma (ESCC)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Principal Investigator, Jun wang, Study Principal Investigator, Hebei Medical University Fourth Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-EC-II-024
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Locally Advanced Unresectable Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Induction stage：Adebrelimab+TC； Treatment stage: TC/PF+ radiation therapy； Maintenance stage: Adebrelimab
  Interventions: Drug: Induction stage：Adebrelimab+TC；Treatment stage: TC/PF+ radiation therapy；Maintenance stage: Adebrelimab

INTERVENTIONS:
Drug: Induction stage：Adebrelimab+TC；Treatment stage: TC/PF+ radiation therapy；Maintenance stage: Adebrelimab — Induction stage：Adebrelimab+TC： Adebrelimab : 1200mg d1, iv, q3w ； TC : paclitaxel 135mg/m2, or nab-paclitaxel paclitaxel 180mg/m2, d1, iv，carboplatin AUC=5, d1, iv, q3w，2 cycles.
  Treatment stage: TC/PF+ radiation therapy:
  PET-CT responders (SUV (PETr) reduction ≥35%)：
  TC/PF+ radiation therapy:
  TC : paclitaxel 50mg/m2, nab-paclitaxel paclitaxel 60mg/m2, d1, iv; carboplatin AUC=2, d1, iv, qw，5 cycles.
  PF : fluorouracil 750-1000mg/m2, CIV 96 hours，cisplatin 75mg/m2, d1, iv, q4w，2 cycles.
  Radiation therapy: 50.4Gy-60Gy/28-33f.
  PET-CT non-responders (SUV (PETr) reduction <35%)：(switch to a different chemotherapy drug which not used during the earlier induction phase)
  PF/TC+ radiation therapy:
  dose same as above.
  Maintenance stage: Adebrelimab:
  Adebrelimab: 1200mg d1, iv, q3w , until disease progression or unacceptable toxicity occurs（Up to one year）.

SUMMARY:
This study aims to evaluate the efficacy and safety of induction Adebrelimab (anti-PD-L1 antibody) combined with chemotherapy, then guided by PET-CT or RECIST1.1 assessment to change the following chemoradiotherapy regiment for locally advanced unresectable ESCC.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-75 years old, both men and women; 2. Histopathology confirmed esophageal squamous cell carcinoma, locally advanced: T1N+M0, T2-4bNxM0; 3. The surgeon assesses that surgery is not feasible or the patient refuses surgical treatment; 4. If technically feasible, all patients are recommended to have local staging determined by endoscopic ultrasound (EUS); The endoscopic examination report or gastrointestinal (GI) clinical records should clearly indicate the T and N stages; Perform PET-CT examination; 5. Except for basal or squamous cell skin cancer, bladder cancer in situ or cervical cancer, there is no history of malignant tumor within 5 years; Patients with malignant tumors who have undergone surgical treatment in the past and those who have survived disease-free for more than 5 years meet the inclusion criteria; 6. Have not received any systemic anti-tumor treatment in the past (systemic chemotherapy, radiotherapy, targeted therapy, immunotherapy, etc.) 7. At least one measurable lesion（According to RECIST 1.1：The long diameter of the measurable lesion on CT scan is ≥10 mm or the short diameter of the enlarged lymph node is ≥15 mm）; 8. ECOG: 0~1; 9. Expected survival period ≥ 12 weeks; 10. Major organ function has to meet the following certeria: (1) Blood routine examination: 1. HB≥90g/L; 2. ANC ≥ 1.5 × 109 / L; 3. PLT ≥ 100 × 109 / L; (2) Biochemical examination: a. ALT and AST < 2.5XULN; b. TBIL ≤ 1.5XULN; c. Cr ≤ 1.5XULN; 11. Left ventricular ejection fraction (LVEF) ≥50%; 12. Female subjects of childbearing age or male who undergo non-surgical sterilization must agree to use at least one medically approved contraceptive measure (such as intrauterine device, contraceptive pill) for contraception during the study treatment period and within 3 months after the end of the study treatment period. For female subjects of childbearing age who undergo non-surgical sterilization, the serum HCG test must be negative within 7 days before the first administration. 13. Participants were willing to join in this study, and written informed consent, good adherence, cooperate with the follow-up.

Exclusion Criteria:

* 1. Previous history of esophageal cancer surgery； 2. Higher risk of esophageal perforation or fistula； 3. Received systemic immunosuppressive therapy within 14 days prior to the first study medication； 4. Known or suspected to have interstitial pneumonia; Other moderate to severe lung diseases that may seriously affect respiratory function; 5. The patient has any active autoimmune disease or history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, enteritis, systemic lupus erythematosus, rheumatoid arthritis; patients with vitiligo, Asthma has been completely relieved in childhood, and patients who do not need any intervention after adulthood can be included; asthma patients who require bronchodilators for medical intervention cannot be included); 6. Human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS), active hepatitis B (HBV DNA ≥ 1000 copies/ml or 500IU/ml), hepatitis C (positive hepatitis C antibody, and HCV-RNA is higher than the lower limit of detection of the analytical method)； 7. Within 6 months, cerebral vascular accidents (including transient ischemic attacks or symptomatic pulmonary embolism) occur; 8. History of cardiovascular disease with significant clinical significance, including but not limited to: (1) congestive heart failure (NYHA grade>2); (2) Unstable angina pectoris; (3) Have experienced myocardial infarction within 3 months; (4) Any supraventricular arrhythmias or ventricular arrhythmias that require treatment or intervention; 9. Severe infections within 4 weeks before study drug administration, or active infection with CTCAE ≥ 2 grade treated with antibiotics within 2 weeks before study drug administration; 10. History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation; 11. History of psychiatric drugs abuse and can't quit or patients with mental disorders; 12. The researchers think inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2025-08-10 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
1-year Progression-Free-Survival (PFS) rate | 12 months
  PFS defined as the time from the date of treatment to the first evidence of disease progression as defined by response evaluation criteria in solid tumors (RECIST) v1.1 or death from any cause.

SECONDARY OUTCOMES:
cCR rate | 12 months
  A clinical complete response rate (cCR) is defined as the complete disappearance of tumor lesions.
Objective Response Rate, ORR | 12 months
  Defined as the proportion of patients who achieved complete response (CR) and partial response (PR) according to RECIST v1.1.
Disease Control Rate, DCR | 12 months
  Defined as the proportion of patients who achieved complete response (CR), partial response (PR), and stable disease (SD) according to RECIST v1.1.
Duration of Response, DoR | 12 months
  Defined as the time from response(when CR or PR is first diagnosed) to disease progression or death due to any cause.
Progression free Survival, PFS | 24 months
  PFS defined as the time from the date of treatment to the first evidence of disease progression as defined by response evaluation criteria in solid tumors (RECIST) v1.1 or death from any cause.
Overall survival, OS | 24 months
  Defined as the time between signing the informed consent form to death due to various causes.
Incidence of adverse events | 24 months
  Use NCI-CTCAE version 5.0 for classification and grading.

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China